CLINICAL TRIAL: NCT02173522
Title: Phase II Open Label Investigation of the Safety and Efficacy of Pre-Operative Prostate Artery Embolization (PAE) Before Radical Prostatectomy in Prostate Cancer Patients
Brief Title: Phase II Investigation of Prostate Artery Embolization (PAE) Before Radical Prostatectomy in Prostate Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Shivank Bhatia (Other)
Collaborators: Merit Medical Systems, Inc. (Industry); Society of Interventional Radiology Foundation (Other)
Responsible Party: Sponsor-Investigator, Shivank Bhatia, Assistant Professor of Clinical Radiology, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20131034
Record Dates: First submitted 2014-05-22; First posted 2014-06-25 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate artery embolization; Robot-assisted laparoscopic radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate artery embolization (PAE) (Experimental): 10 patients will receive prostate artery embolization (PAE) prior to robot-assisted laparoscopic radical prostatectomy (RALRP).
  Interventions: Device: Prostate artery embolization (PAE)
- Control (No Intervention): 10 patients, matched to PAE patients by risk score, will receive RALRP without PAE. RALRP without PAE is the current standard of care treatment for prostate cancer at the Sylvester Comprehensive Cancer Center.

INTERVENTIONS:
Device: Prostate artery embolization (PAE) — Embolization of the arteries carrying blood to the prostate. All PAE procedures will be conducted with Embosphere Microspheres.
  Arms: Prostate artery embolization (PAE)

SUMMARY:
The purpose of this study is to determine whether pre-operative prostate artery embolization (PAE) reduces intra-operative blood loss and improves surgical outcomes among prostate cancer patients undergoing robot-assisted laparoscopic radical prostatectomy (RALRP).

DETAILED DESCRIPTION:
Duration of study:

This study will enroll 20 patients, with a target enrollment period of 18 months. Patients who undergo prostate artery embolization (PAE) will have follow-up visits 2 weeks and 6 weeks after PAE. All patients in the study will have post RALRP follow-up visits at 2 weeks, 3 months, 6 months, 9 months, and 12 months after surgery. All patients will continue to be followed according to the usual standard of care following the completion of the study.

Study design:

The first 10 patients who meet all study eligibility criteria and provide consent for participation in the study will receive PAE prior to RALRP. Control patients will be matched 1:1 to PAE patients, according to risk score, and will receive RALRP without PAE. Control patients will be selected after all PAE patients have been enrolled, and need not meet all study eligibility criteria.

The following assessments and evaluations are required for participation in this study:

Physical exams, blood & urine tests, magnetic resonance imaging (MRI), digital rectal exams (DREs), transrectal ultrasound (TRUS), Expanded Prostate Cancer Index Composite (EPIC) questionnaires, International Index of Erectile Function (IIEF) questionnaires, robot-assisted laparoscopic radical prostatectomy (RALRP), and pad weight tests. All patients enrolled in the PAE arm of the study will undergo embolization of the blood vessels that feed the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 45-79 years old
* Patient has signed informed consent
* Patient has biopsy-proven prostate adenocarcinoma with localized disease
* Patient is a candidate for robot-assisted laparoscopic radical prostatectomy (RALRP)
* Patient has a prostate size >40 grams

Exclusion Criteria:

* Active urinary tract infection
* History of life threatening allergy to iodinated contrast agents
* Any known condition that limits catheter-based intervention or is a contraindication to embolization (eg shunt or adverse arterial anatomy)
* Patient is unable to undergo MRI imaging
* Cardiac condition including congestive heart failure or uncontrolled arrhythmia, uncontrolled diabetes mellitus, significant respiratory disease, or known immunosuppression which required hospitalization within the previous 6 months
* Baseline serum creatinine level > 1.8 mg/dL
* Baseline hemoglobin < 8.0 g/dL
* Active cystolithiasis or prostatitis
* History of pelvic irradiation or radical pelvic surgery
* Known major iliac arterial occlusive disease
* Confirmed or suspected bladder cancer
* Urethral strictures, bladder neck contracture, or other bladder or urethral pathology that could limit catheterization
* Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease if the therapy or patient evaluation may potentially cause injury to sites of previous rectal surgery, e.g. if a transrectal probe is used
* Previous pelvic irradiation or radical pelvic surgery
* Previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate
* Prior transurethral resection of the prostate or other invasive therapies
* Coagulation disturbances not normalized by medical treatment
* Acute urinary retention
* Hypersensitivity to gelatin products
* Any contraindication to embolization, including intolerance to vessel occlusion procedures, vascular anatomy/blood flow that precludes catheter placement or embolic agent injection, presence/likely onset of vasospasm, presence/likely onset of hemorrhage, severe atheromatous disease, feeding arteries smaller than distal branches, arteriovenous shunt, and collateral vessel pathways endangering normal territories during embolization or pelvic inflammatory disease

Ages: 45 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivank Bhatia, MD, Principal Investigator — University of Miami
Locations (1):
- Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prostate Artery Embolization (PAE) | Control
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: subject analyzed in PAE arm 4. 0 subject analyzed in the control arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Artery Embolization (PAE) | Control | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 0 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss During Robot-assisted Laparoscopic Radical Prostatectomy (RALRP)
Description: Blood loss during the robotic prostatectomy will be estimated by the surgeon performing the procedure.
Time Frame: RALRP procedure, up to 3 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
mL | 110 (10)

2. Secondary Outcome: Change in Hemoglobin Compared to Baseline
Description: Patients will undergo a blood test to assess their hemoglobin level prior to surgery on the day of RALRP, and again on post operative day 1 to determine the change in the hemoglobin level following surgery.
Time Frame: Baseline, RALRP post operative day
Measure: Mean (Standard Deviation); unit: G/DL
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
G/DL
  BASELINE | 14.3 (0.725)
  POST RALRP DAY 1 | 11.77 (1.33)

3. Secondary Outcome: Change in Hematocrit
Description: Patients will undergo a blood test to assess their hematocrit prior to surgery on the day of RALRP, and again on post operative day 1 to determine the change in the hematocrit following surgery.
Time Frame: Baseline, RALRP post operative day 1
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
percentage of red blood cells
  BASELINE | 39.65 (1.99)
  POST RALRP DAY 1 | 36.92 (1.63)

4. Secondary Outcome: Change in Prostate Volume
Description: Patients who receive PAE will undergo MRIs before PAE and 6 weeks after PAE to assess any change in prostate volume following the embolization procedure.
Time Frame: Baseline, 6 weeks post PAE
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
cc
  Baseline | 124.6 (30.54)
  Week 6 | 91.55 (32.13)

5. Secondary Outcome: Number of Patients That Required Blood Transfusion
Description: Requirement for blood transfusion during the prostatectomy procedure will be assessed in all patients. The surgeon performing the prostatectomy will determine whether or not patients require blood transfusions.
Time Frame: RALRP procedure
Measure: Number; unit: participants
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
participants | 0

6. Secondary Outcome: RALRP Duration
Time Frame: RALRP procedure
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
hr | 2.5 (1.15)

7. Secondary Outcome: Length of Hospital Stay After RALRP
Time Frame: 48 hours post procedure
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
Days | 2 (0.43)

8. Secondary Outcome: Number of Participants for Whom Prostatectomy Procedure Did Not Succeed in Removing the Entire Cancer
Description: Histopathology examination post RALRP will be used to determine if the prostatectomy procedure succeeded in removing the entire cancer.
Time Frame: RALRP procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
Participants | 4

9. Secondary Outcome: Biochemical Recurrence of Prostate Cancer
Description: Biochemical recurrence of prostate cancer will be determined by PSA levels 1 year following the RALRP procedure.
Time Frame: 1 year post RALRP
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
ng/mL | 0.067 (0.0427)

10. Secondary Outcome: Return to Continence
Description: Return to continence following the RALRP procedure will be determined by the pad weight test, conducted at each follow-up visit until the patient is continent.
Time Frame: An expected average of 1 week post RALRP
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
grams | 463 (496.50)

11. Secondary Outcome: RALRP-related Adverse Events
Description: Any adverse event occurring between the date of RALRP and 1 year of follow-up that the investigators determine to be related to the RALRP procedure will be assessed.
Time Frame: Through 1 year post RALRP
Measure: Number; unit: adverse events
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
adverse events | 4

12. Secondary Outcome: PAE-related Adverse Events
Description: Any adverse event occurring between the date of PAE and 1 year of follow-up that the investigators determine to be related to the PAE procedure will be assessed.
Time Frame: Through 1 year post RALRP
Measure: Number; unit: adverse events
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
adverse events | 9

13. Secondary Outcome: Change From Baseline in Erectile Function at One Year Post RALRP
Description: The International Index of Erectile Function (IIEF) questionnaire is a multi-dimensional self-administered test found to be used in the clinical assessment of erectile dysfunction. It examines the 4 main domains of male sexual function. A higher score would indicated less dysfunction. The scores can range 6 to 75
Time Frame: Baseline,1 year post RALRP
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
Score on a scale | 17 (8.286)

14. Secondary Outcome: Change in PSA Following PAE
Description: Patients who undergo PAE will have blood tests to determine the change in their PSA levels between baseline and 6 weeks post PAE.
Time Frame: 6 weeks post PAE
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
ng/mL
  baseline | 9.9125 (5.22)
  week 6 | 5.94 (5.06)

15. Secondary Outcome: Histologic Changes in the Prostate After PAE
Description: The Gleason Score prostate Cancer Grading and Prognostic scoring system will be used to determine the histologic changes in the prostate tumor. Since prostate tumors are often made up of cancerous cells that have different grades, two grades are assigned to each patient. A primary grade is given to describe the cells that make up the largest area of the tumor and a secondary grade is given to describe the cells of the next largest area. The sums of the scores will be evaluated. The Gleason Score sum will range from 1 - 10, with the higher score indicating a more advanced neoplasm.
Time Frame: Between baseline prostate biopsy and RALRP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prostate Artery Embolization (PAE)
Number analyzed (Participants) | 4
Units on a scale
  Baseline | 5.25 (3.5)
  Post RALP | 3.75 (3.77)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Prostate Artery Embolization (PAE)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prostate Artery Embolization (PAE) (N=4)
Ventricular Arrhythmia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prostate Artery Embolization (PAE) (N=4)
Hematuria (Renal and urinary disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 2
Cystitis (Renal and urinary disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Bladder Spasm (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Flu Like Symptoms (General disorders) | 1
Nausea (Nervous system disorders) | 1
Edema Limbs (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Wound Complication (Infections and infestations) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Acute Kidney injury (Renal and urinary disorders) | 1
Creatinine increased (Investigations) | 1
Hematoma (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT02173522/Prot_SAP_000.pdf